CLINICAL TRIAL: NCT04015804
Title: European Ambispective Cohort of Rectal Cancer Patient Who Underwent Robotic Low Anterior Resection
Brief Title: Robotic Low Rectum Anterior Resection
Acronym: GROG-R01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICM-BDD 2015/05
Record Dates: First submitted 2019-07-04; First posted 2019-07-11 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Rectum Cancer
Keywords: cancer; rectum; robot
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical database (Other)
  Interventions: Other: Clinical database

INTERVENTIONS:
Other: Clinical database — Creation of an ambispective (retrospective and prospective), multicentric and European clinical database for surgery with robotic assistance in rectal cancers with implementation in France and then in Europe

SUMMARY:
The laparoscopic approach for total mesorectal excision (L-TME) results improved short-term outcomes. However this approach has technical limitations when the pelvis is narrow and deep. Indeed there is a limited mobility of straight laparoscopic instruments and associated loss of dexterity, unstable camera view and compromised ergonomics for the surgeon. Robotic technology was developed to reduce these limitations and offers the advantages of intuitive manipulation of laparoscopic instruments with wrist articulation, a 3-dimensional field of view, a stable camera platform with zoom magnification, dexterity enhancement and an ergonomic operating environment. A major advantage of the robotic approach is the surgeon's simultaneous control of the camera and of the two or three additional instruments. This advantage facilitates traction and counter-traction. The technological advantages of robotic surgery should also allow a finer dissection in a narrow pelvic cavity.

DETAILED DESCRIPTION:
The laparoscopic approach for laparoscopic total mesorectal excision (L-TME) results improved short-term outcomes and provides a clearer intraoperative view compared with the open approach in a deep and narrow pelvis. Preliminary results from the COLOR II trial confirmed improved patient recovery and similar safety, same resection margins and completeness of resection using L-TME compared with the results achieved with open surgery.Results from the CLASICC trial supported the use of laparoscopic surgery for colorectal cancer and showed no difference between laparoscopically-assisted TME and conventional open resection at 10 years post-procedure in terms of overall survival, disease-free survival and local recurrence.

Despite these positive clinical outcomes for L-TME, laparoscopic resection of rectal cancer, especially in a deep and narrow pelvis, is technically demanding and demands a long learning curve. Technical limitations include limited mobility of straight laparoscopic instruments and associated loss of dexterity, unstable camera view and compromised ergonomics for the surgeon. These limitations could explain the conversion rate which remained at 17% in the last COLOR II trial.2 In order to avoid this drawback, we have described for patients with high-risk of conversion, the trans-anal endoscopic proctectomy (TAEP) approach performed with the Transanal Endoscopic Operation (TEO) device.This trans-anal procedure is also called trans anal minimally invasive surgery (TAMIS) if a laparoscopic port is used.

Robotic technology was developed to reduce these limitations and offers the advantages of intuitive manipulation of laparoscopic instruments with wrist articulation, a 3-dimensional field of view, a stable camera platform with zoom magnification, dexterity enhancement and an ergonomic operating environment. A major advantage of the robotic approach is the surgeon's simultaneous control of the camera and of the two or three additional instruments. This advantage facilitates traction and counter-traction. The technological advantages of robotic surgery should also allow a finer dissection in a narrow pelvic cavity. However, total robotic surgery for rectal cancer is still technically challenging and involves two operative fields (splenic flexure and rectum), potential collision of the robotic arms and lack of tactile feedback.

Reports of robotic and laparoscopic rectal cancer surgery outcomes showed similar intraoperative results and morbidity, postoperative recovery and short-term oncologic outcomes.However, longer operation times have been described as a disadvantage of the robotic system, compared with conventional laparoscopy. On the other hand, all meta-analyses comparing robotic total mesorectal excision (R-TME) and L-TME concluded in reduction of the conversion rate.

Since 2007, the rectal surgery with robotic assistance is booming. To date, seven meta-analyzes have been published. All show that the robot exceeds laparoscopy to reduce the conversion rate. The last two meta-analyzes that had gathered more than 800 patients undergoing robotic surgery have again highlighted the contribution of the robot to secure the radial margin and decrease sexual sequelae. However, there is not so far from Phase 3 randomized trial dealing with the subject. The ROLARR protocol was completed in late 2014 (Ph III laparoscopy / Robot), the first results are published in late 2015.

The interest of a European multicenter ambispective (retrospective and prospective) database is fundamental because this early work suggests that the robot can make more for specific subgroups of patients, particularly in high surgical risk patients (Male, narrow pelvis, high BMI, mesorectal fat, large tumor of the anterior and middle third).

The largest series of R-TME stems from the US national cancer database (965 patients operated by R-TME) and confirms a 9.5% conversion rate compared to 16.4% with L-TME (p < 0.001).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 years
2. Introducing rectal cancer, colorectal junction eligible to robotic surgery support from June 2015
3. Treatment Naive for this cancer
4. Enjoying a social protection scheme (For France only)
5. Patient followed in the participant center

Exclusion Criteria:

1. Male or female age (s) under 18 years
2. Private person of liberty or under supervision (including guardianship)
3. People who do not speak French (For France only)
4. Major Nobody unable to consent
5. Patient GROG-R01 already included in the base
6. Patient Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Conversion rate for robotic surgery | 5 years

SECONDARY OUTCOMES:
Anatomo-pathological curability criteria | 5 years
Median of hospitalization time | 5 years
Post-operative morbidity | 5 years
Number of robot docking | 5 years
Operating time | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Rouanet, MD, Study Chair — Institut régional du cancer de Montpellier
Locations (19):
- UCL, Brussels, Belgium
- France (17):
  - Hôpital Européen, Marseille, Bouches Du Rhône
  - Institut Paoli Calmettes, Marseille, Bouches Du Rhône
  - Centre François Baclesse, Caen, Calvados
  - Clinique Kennedy, Nîmes, Gard
  - Clinique Saint Jean du Languedoc, Toulouse, Haute Garonne
  - CHU Dupuytren, Limoges, Haute Vienne
  - Hôpital privé d'Anthony, Antony, Hauts De Seine
  - Institut régional du cancer de Montpellier, Montpellier, Hérault
  - Hôpital Michalon, Grenoble, Isère
  - CHU de Nantes, Nantes, Loire Atlantique
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Loire Atlantique
  - CHR Orléans, Orléans, Loiret
  - CHU de Nancy, Vandœuvre-lès-Nancy, Lorraine
  - Centre Oscart Lambret, Lille, Nord
  - Institut Gustave Roussy, Villejuif, Val De Marne
  - Hôpital Diaconesses, Paris
  - Hôpital européen Georges Pompidou, Paris
- Centre Hospitalier-Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Green BL, Marshall HC, Collinson F, Quirke P, Guillou P, Jayne DG, Brown JM. Long-term follow-up of the Medical Research Council CLASICC trial of conventional versus laparoscopically assisted resection in colorectal cancer. Br J Surg. 2013 Jan;100(1):75-82. doi: 10.1002/bjs.8945. Epub 2012 Nov 6. PMID 23132548
- [Background] van der Pas MH, Haglind E, Cuesta MA, Furst A, Lacy AM, Hop WC, Bonjer HJ; COlorectal cancer Laparoscopic or Open Resection II (COLOR II) Study Group. Laparoscopic versus open surgery for rectal cancer (COLOR II): short-term outcomes of a randomised, phase 3 trial. Lancet Oncol. 2013 Mar;14(3):210-8. doi: 10.1016/S1470-2045(13)70016-0. Epub 2013 Feb 6. PMID 23395398
- [Background] Rouanet P, Mourregot A, Azar CC, Carrere S, Gutowski M, Quenet F, Saint-Aubert B, Colombo PE. Transanal endoscopic proctectomy: an innovative procedure for difficult resection of rectal tumors in men with narrow pelvis. Dis Colon Rectum. 2013 Apr;56(4):408-15. doi: 10.1097/DCR.0b013e3182756fa0. PMID 23478607
- [Background] Fernandez-Hevia M, Delgado S, Castells A, Tasende M, Momblan D, Diaz del Gobbo G, DeLacy B, Balust J, Lacy AM. Transanal total mesorectal excision in rectal cancer: short-term outcomes in comparison with laparoscopic surgery. Ann Surg. 2015 Feb;261(2):221-7. doi: 10.1097/SLA.0000000000000865. PMID 25185463
- [Background] Sylla P, Rattner DW, Delgado S, Lacy AM. NOTES transanal rectal cancer resection using transanal endoscopic microsurgery and laparoscopic assistance. Surg Endosc. 2010 May;24(5):1205-10. doi: 10.1007/s00464-010-0965-6. Epub 2010 Feb 26. PMID 20186432
- [Background] Atallah S, Martin-Perez B, Albert M, deBeche-Adams T, Nassif G, Hunter L, Larach S. Transanal minimally invasive surgery for total mesorectal excision (TAMIS-TME): results and experience with the first 20 patients undergoing curative-intent rectal cancer surgery at a single institution. Tech Coloproctol. 2014 May;18(5):473-80. doi: 10.1007/s10151-013-1095-7. Epub 2013 Nov 23. PMID 24272607
- [Background] D'Annibale A, Pernazza G, Monsellato I, Pende V, Lucandri G, Mazzocchi P, Alfano G. Total mesorectal excision: a comparison of oncological and functional outcomes between robotic and laparoscopic surgery for rectal cancer. Surg Endosc. 2013 Jun;27(6):1887-95. doi: 10.1007/s00464-012-2731-4. Epub 2013 Jan 5. PMID 23292566
- [Background] Kwak JM, Kim SH, Kim J, Son DN, Baek SJ, Cho JS. Robotic vs laparoscopic resection of rectal cancer: short-term outcomes of a case-control study. Dis Colon Rectum. 2011 Feb;54(2):151-6. doi: 10.1007/DCR.0b013e3181fec4fd. PMID 21228661
- [Background] Park JS, Choi GS, Lim KH, Jang YS, Jun SH. Robotic-assisted versus laparoscopic surgery for low rectal cancer: case-matched analysis of short-term outcomes. Ann Surg Oncol. 2010 Dec;17(12):3195-202. doi: 10.1245/s10434-010-1162-5. Epub 2010 Jun 30. PMID 20589436
- [Background] Patel CB, Ragupathi M, Ramos-Valadez DI, Haas EM. A three-arm (laparoscopic, hand-assisted, and robotic) matched-case analysis of intraoperative and postoperative outcomes in minimally invasive colorectal surgery. Dis Colon Rectum. 2011 Feb;54(2):144-50. doi: 10.1007/DCR.0b013e3181fec377. PMID 21228660
- [Background] Bianchi PP, Ceriani C, Locatelli A, Spinoglio G, Zampino MG, Sonzogni A, Crosta C, Andreoni B. Robotic versus laparoscopic total mesorectal excision for rectal cancer: a comparative analysis of oncological safety and short-term outcomes. Surg Endosc. 2010 Nov;24(11):2888-94. doi: 10.1007/s00464-010-1134-7. Epub 2010 Jun 5. PMID 20526623
- [Background] Popescu I, Vasilescu C, Tomulescu V, Vasile S, Sgarbura O. The minimally invasive approach, laparoscopic and robotic, in rectal resection for cancer. A single center experience. Acta Chir Iugosl. 2010;57(3):29-35. doi: 10.2298/aci1003029p. PMID 21066980
- [Background] Lin S, Jiang HG, Chen ZH, Zhou SY, Liu XS, Yu JR. Meta-analysis of robotic and laparoscopic surgery for treatment of rectal cancer. World J Gastroenterol. 2011 Dec 21;17(47):5214-20. doi: 10.3748/wjg.v17.i47.5214. PMID 22215947
- [Background] Trastulli S, Farinella E, Cirocchi R, Cavaliere D, Avenia N, Sciannameo F, Gulla N, Noya G, Boselli C. Robotic resection compared with laparoscopic rectal resection for cancer: systematic review and meta-analysis of short-term outcome. Colorectal Dis. 2012 Apr;14(4):e134-56. doi: 10.1111/j.1463-1318.2011.02907.x. PMID 22151033
- [Background] Memon S, Heriot AG, Murphy DG, Bressel M, Lynch AC. Robotic versus laparoscopic proctectomy for rectal cancer: a meta-analysis. Ann Surg Oncol. 2012 Jul;19(7):2095-101. doi: 10.1245/s10434-012-2270-1. Epub 2012 Feb 16. PMID 22350601
- [Background] Yang Y, Wang F, Zhang P, Shi C, Zou Y, Qin H, Ma Y. Robot-assisted versus conventional laparoscopic surgery for colorectal disease, focusing on rectal cancer: a meta-analysis. Ann Surg Oncol. 2012 Nov;19(12):3727-36. doi: 10.1245/s10434-012-2429-9. Epub 2012 Jul 3. PMID 22752371
- [Background] Gonzalez Fernandez AM, Mascarenas Gonzalez JF. [Total laparoscopic mesorectal excision versus robot-assisted in the treatment of rectal cancer: a meta-analysis]. Cir Esp. 2012 Jun-Jul;90(6):348-54. doi: 10.1016/j.ciresp.2012.03.004. Epub 2012 Apr 24. Spanish. PMID 22537895
- [Background] Ortiz-Oshiro E, Sanchez-Egido I, Moreno-Sierra J, Perez CF, Diaz JS, Fernandez-Represa JA. Robotic assistance may reduce conversion to open in rectal carcinoma laparoscopic surgery: systematic review and meta-analysis. Int J Med Robot. 2012 Sep;8(3):360-70. doi: 10.1002/rcs.1426. Epub 2012 Mar 22. PMID 22438060
- [Background] Xiong B, Ma L, Zhang C, Cheng Y. Robotic versus laparoscopic total mesorectal excision for rectal cancer: a meta-analysis. J Surg Res. 2014 May 15;188(2):404-14. doi: 10.1016/j.jss.2014.01.027. Epub 2014 Jan 22. PMID 24565506
- [Background] Son GM, Kim JG, Lee JC, Suh YJ, Cho HM, Lee YS, Lee IK, Chun CS. Multidimensional analysis of the learning curve for laparoscopic rectal cancer surgery. J Laparoendosc Adv Surg Tech A. 2010 Sep;20(7):609-17. doi: 10.1089/lap.2010.0007. PMID 20701545
- [Background] Kim HJ, Choi GS, Park JS, Park SY. Multidimensional analysis of the learning curve for robotic total mesorectal excision for rectal cancer: lessons from a single surgeon's experience. Dis Colon Rectum. 2014 Sep;57(9):1066-74. doi: 10.1097/DCR.0000000000000174. PMID 25101602
- [Background] Jimenez-Rodriguez RM, Diaz-Pavon JM, de la Portilla de Juan F, Prendes-Sillero E, Dussort HC, Padillo J. Learning curve for robotic-assisted laparoscopic rectal cancer surgery. Int J Colorectal Dis. 2013 Jun;28(6):815-21. doi: 10.1007/s00384-012-1620-6. Epub 2012 Dec 15. PMID 23242270
- [Background] Kuo LJ, Lin YK, Chang CC, Tai CJ, Chiou JF, Chang YJ. Clinical outcomes of robot-assisted intersphincteric resection for low rectal cancer: comparison with conventional laparoscopy and multifactorial analysis of the learning curve for robotic surgery. Int J Colorectal Dis. 2014 May;29(5):555-62. doi: 10.1007/s00384-014-1841-y. Epub 2014 Feb 23. PMID 24562546
- [Background] Baek JH, Pastor C, Pigazzi A. Robotic and laparoscopic total mesorectal excision for rectal cancer: a case-matched study. Surg Endosc. 2011 Feb;25(2):521-5. doi: 10.1007/s00464-010-1204-x. Epub 2010 Jul 7. PMID 20607559
- [Background] Park YA, Kim JM, Kim SA, Min BS, Kim NK, Sohn SK, Lee KY. Totally robotic surgery for rectal cancer: from splenic flexure to pelvic floor in one setup. Surg Endosc. 2010 Mar;24(3):715-20. doi: 10.1007/s00464-009-0656-3. Epub 2009 Aug 18. PMID 19688388
- [Background] Speicher PJ, Englum BR, Ganapathi AM, Nussbaum DP, Mantyh CR, Migaly J. Robotic Low Anterior Resection for Rectal Cancer: A National Perspective on Short-term Oncologic Outcomes. Ann Surg. 2015 Dec;262(6):1040-5. doi: 10.1097/SLA.0000000000001017. PMID 25405559
- [Background] Tuech JJ, Karoui M, Lelong B, De Chaisemartin C, Bridoux V, Manceau G, Delpero JR, Hanoun L, Michot F. A step toward NOTES total mesorectal excision for rectal cancer: endoscopic transanal proctectomy. Ann Surg. 2015 Feb;261(2):228-33. doi: 10.1097/SLA.0000000000000994. PMID 25361216
- [Background] Wolthuis AM, de Buck van Overstraeten A, D'Hoore A. Dynamic article: transanal rectal excision: a pilot study. Dis Colon Rectum. 2014 Jan;57(1):105-9. doi: 10.1097/DCR.0000000000000008. PMID 24316953
- [Background] Dumont F, Goere D, Honore C, Elias D. Transanal endoscopic total mesorectal excision combined with single-port laparoscopy. Dis Colon Rectum. 2012 Sep;55(9):996-1001. doi: 10.1097/DCR.0b013e318260d3a0. PMID 22874608
- [Background] Zorron R, Phillips HN, Coelho D, Flach L, Lemos FB, Vassallo RC. Perirectal NOTES access: "down-to-up" total mesorectal excision for rectal cancer. Surg Innov. 2012 Mar;19(1):11-9. doi: 10.1177/1553350611409956. Epub 2011 Jul 7. PMID 21742663